CLINICAL TRIAL: NCT01629485
Title: Part vs Whole Task Mastery Simulation Training for Laparoscopic Hernia Repair: A Randomized Trial
Brief Title: Part vs Whole Task Mastery Training for Laparoscopic Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David R. Farley, Co-Director of the Mayo Simulation Center, Professor of Surgery, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11-005712
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Hernia
Keywords: Mastery Learning; Surgical Education; Laparoscopic Hernia Repair; Part vs Whole Task; Contextual Interference; laparoscopy; training; curriculum
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole Task (Experimental): Trainees will undergo whole task mastery training in the TEP simulator after completing the video curriculum portion.
  Interventions: Behavioral: Online Video Curriculum; Behavioral: Whole Task Mastery Training
- Part Task (Experimental): Trainees will undergo a random part task mastery training in the TEP simulator after completing the video portion of the curriculum.
  Interventions: Behavioral: Online Video Curriculum; Behavioral: Part Task Mastery Training

INTERVENTIONS:
Behavioral: Online Video Curriculum — A video curriculum has been designed for the purpose of educating general surgery residents in laparoscopic hernia repairs. The curriculum covers topics from basic anatomy, selection of patients, management, and operative technique.
Behavioral: Whole Task Mastery Training — Trainees will undergo whole task mastery training in the TEP simulator. The benchmarks for mastery training in the setting of whole task tep repairs was established with performance measures of multiple staff surgeons previously.
  Arms: Whole Task
Behavioral: Part Task Mastery Training — Trainees will undergo part task mastery training in the TEP simulator. The benchmarks for mastery training in the setting of part task tep repairs was established with performance measures of multiple staff surgeons previously.
  Arms: Part Task

SUMMARY:
The investigators will perform a randomized controlled trial with a stratified-block design to compare the effect of the part versus whole task simulation training for TEP repairs.

ELIGIBILITY:
Inclusion Criteria:

* Study Participants: Only residents who have achieved mastery of the TEP training curriculum (in either arm) will be eligible for OR assessment
* Patients: All patients deemed fit by the staff supervising surgeon to undergo a TEP repair will be considered for this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Operative Time | Measured in Seconds
  Operative Time will be measured with a chronometer. Staff take overs and down time will be excluded from the trainee's time. Trainee time will be defined as when he/she has the instruments in his/her hands and is actively doing the case.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Hernandez-Irizarry, BS, Principal Investigator — Mayo Clinic; David Farley, MD, Principal Investigator — Mayo Clinic; Benjamin Zendejas, MD/MsC, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States